CLINICAL TRIAL: NCT06716814
Title: A Multinational, Prospective, Open-label, Roll-over Study (LIBERTY) to Provide Post-trial Access to Treatment for Patients With Severe Haemophilia A Who Have Completed a Previous Trial With Efanesoctocog Alfa
Brief Title: Study to Provide Continued Access to Treatment for Patients Completing a Previous Trial With Efanesoctocog Alfa
Acronym: LIBERTY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.BIVV001-002; 2023-506537-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-02; First posted 2024-12-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Severe Haemophilia A
Keywords: Haemophilia A; Blood coagulation disorder; Factor VIII; FVIII; Coagulation protein disorder; Severe Haemophilia A; Efanesoctocog alfa
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Coagulation Protein Disorders | interventions — BIVV001

STUDY DESIGN:
Intervention Model Description: Roll-over study to provide post-trial access to treatment for patients with severe haemophilia A who have completed a previous trial with efanesoctocog alfa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Efanesoctocog alfa phrophylaxis (Experimental): Patients who have completed a previous study with efanesoctocog alfa may continue to be treated with a prophylactic dose of 50 IU/kg efanesoctocog alfa once weekly.
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — Treatment starts when the patient completes the parent study and continues until efanesoctocog alfa is commercially available in each patient's respective country, or until March 2027, whichever comes first.
  Other Names: BIVV001; Altuvoct; Altuviiio; Recombinant coagulation factor VIII Fc-von-Willebrand Factor-XTEN fusion protein (rFVIIIFc-VWF-XTEN)

SUMMARY:
This is a multinational, prospective, open-label, roll-over study in patients with severe haemophilia A, ≥6 years of age, who have completed participation in any of the parental studies with efanesoctocog alfa; XTEND-ed study (LTS16294), FREEDOM study (Sobi.BIVV001-001), or PK comparison study (Sobi.BIVV001-003). The aim of the study is to provide patients with continuous benefit from efanesoctocog alfa treatment and to further continue clinical monitoring for safety and efficacy until efanesoctocog alfa is commercially available in each patient's respective country (or until March 2027, whichever comes first).

The study starts with the Baseline Visit, which will be done in connection to the End of Study visit (or equivalent) in the respective parent study. Subsequent study visits (on site or phone call) will be done approximately every 13 weeks until End of Treatment. An End of Study safety phone call will be done 14 (+7) days after the End of Treatment Visit.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent. Parents or legally designated representatives' consent is required for patients who are below 18 years of age or unable to give consent. Patients who are below 18 years of age may provide assent in addition to the parents'/legally designated representatives' consent, if appropriate.
* Must have completed one of the required parent studies: Sobi.BIVV001-001, Sobi.BIVV001-003, or LTS16294, and be receiving a clinical benefit from the efanesoctocog alfa treatment, as judged by the Investigator.
* Willingness and ability of patient or their parent or legally designated representative to complete training in the use of the study patient diary and to complete the diary throughout the study.

Exclusion Criteria:

* Positive inhibitor result (assessed by central laboratory), defined as ≥0.6 Bethesda units (BU)/mL, at Baseline Visit.
* Ongoing or planned participation in any interventional clinical study at Baseline Visit.
* Patient not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of injections to treat a bleeding episode | From enrollment and up to 52 weeks
Total dose to treat a bleeding episode | From enrollment and up to 52 weeks
Adverse events (AEs), including serious adverse events (SAEs) and adverse events of special interest (AESIs) | From enrollment and up to 52 weeks
  Number of participants with occurrence of AEs, SAEs, and AESIs
Annualized bleeding rate (ABR) for treated bleeding episodes | From enrollment and up to 52 weeks
  ABR for treated bleeding episodes during prophylactic treatment.
Annualized bleeding rate (ABR) for treated bleeding episodes by type of bleed | From enrollment and up to 52 weeks
  ABR for treated bleeding episodes during prophylactic treatment by type of bleed.
Annualized bleeding rate (ABR) for treated bleeding episodes by location of bleed | From enrollment and up to 52 weeks
  ABR for treated bleeding episodes during prophylactic treatment by location of bleed.
Annualized bleeding rate (ABR) for all bleeding episodes | From enrollment and up to 52 weeks
  ABR for all bleeding episodes (including untreated bleeding episodes, excluding surgery bleeds) during prophylactic treatment.
Annualized bleeding rate (ABR) for all bleeding episodes by type of bleed | From enrollment and up to 52 weeks
  ABR for all bleeding episodes (including untreated bleeding episodes, excluding surgery bleeds) during prophylactic treatment, by type of bleed.
Annualized bleeding rate (ABR) for all bleeding episodes by location of bleed | From enrollment and up to 52 weeks
  ABR for all bleeding episodes (including untreated bleeding episodes, excluding surgery bleeds) during prophylactic treatment, by location of bleed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Development Lead, Study Director — Sobi AB
Locations (22):
- Bulgaria (2):
  - Sobi Investigational Site, Plovdiv
  - Sobi Investigational Site, Sofia
- France (7):
  - Sobi Investigational Site, Bordeaux
  - Sobi Investigational Site, Brest
  - Sobi Investigational Site, Bron
  - Sobi Investigational Site, Le Kremlin-Bicêtre
  - Sobi Investigational Site, Lille
  - Sobi Investigational Site, Marseille
  - Sobi Investigational Site, Strasbourg
- Sobi Investigational Site, Athens, Greece
- Italy (8):
  - Sobi Investigational Site, Catanzaro
  - Sobi Investigational Site, Florence
  - Sobi Investigational Site, Milan
  - Sobi Investigational Site, Naples
  - Sobi Investigational Site, Parma
  - Sobi Investigational Site, Rome
  - Sobi Investigational Site, Rozzano
  - Sobi Investigational Site, Vicenza
- Sobi Investigational Site, Oslo, Norway
- Spain (2):
  - Sobi Investigational Site, A Coruña
  - Sobi Investigational Site, Zaragoza
- Sobi Investigational Site, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sobi data sharing criteria and process for requesting access can be found at: https:// www.sobi.com/en/policies
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year following completion of the trial, or at the time of CSR finalization.
Access Criteria: A decision on sharing will be based on the following:
  The scientific merit of the proposal - i.e. the proposal should be scientifically sound, ethical, and have the potential to contribute to the advancement of public health. The feasibility of the research proposal - i.e. the requesting research team must be scientifically qualified and have the resources to conduct the proposed project. Maintenance of personal integrity - i.e. Sobi will not consider sharing individual data if there is a risk of re-identification of individuals despite a proper anonymisation. Moreover, the patients' informed consent will always be respected. Sobi reserves the right to reject the proposal if the anonymisation process will render unusable data. Publication of results - the applicants should commit to submit their findings to a peer-reviewed scientific journal, alternatively to present the results at a congress (poster or similar), regardless of the research outcome.
URL: https://www.sobi.com/en/policies